CLINICAL TRIAL: NCT05240339
Title: Characterization and Progression of Minor Phenomena in Parkinson's Disease
Brief Title: Characterization and Progression of Minor Phenomena in Parkinson's Disease (PD)
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Principal Investigator, Ruth Schneider, MD, Associate Professor, University of Rochester
Other Study IDs: STUDY00003440
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease; Parkinson Disease Psychosis; Hallucinations; Delusion
MeSH Terms: conditions — Parkinson Disease; Hallucinations; Delusions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD participants with minor phenomena
  Interventions: Other: Observation of minor phenomena

INTERVENTIONS:
Other: Observation of minor phenomena — observation twice a year over 3 years

SUMMARY:
Parkinson's disease psychosis encompasses a range of symptoms, including minor phenomena, frank hallucinations, and delusions. Minor phenomena include passage hallucinations (fleeting sense of a person, animal or object passing in the periphery), presence hallucinations (feeling of nearby presence), and illusions (misrepresentation of external stimuli). Some forms of PD psychosis may be progressive. The primary objective of this study is to:

1) To determine the cumulative probability of developing hallucinations or delusions over time in individuals with PD minor phenomena followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (as determined by Movement Disorders Society diagnostic criteria for clinically probable Parkinson's disease)
* Parkinson's disease minor phenomena
* ≥30 years of age
* Proficient in English
* Willing and able to provide informed consent

Exclusion Criteria:

* Any current or prior history of formed hallucinations or delusions
* Current or prior treatment with an antipsychotic medication (regardless of indication)
* Diagnosis of mania with psychotic features, bipolar or related disorder, depression with psychotic features, or a psychotic disorder
* Unable or unwilling to complete study activities
* Any medical or psychiatric comorbidity that, in the opinion of the investigator, would compromise study participation

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must meet criteria for clinically probable PD according to the MDS clinical diagnostic criteria for PD. Notably, in these new criteria, PD and dementia with Lewy bodies are recognized as most likely existing on a continuous spectrum and dementia is not an exclusion criterion for PD.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative probability of developing hallucinations or delusions over time | baseline to 36 months
  Kaplan-Meier curves will be used to describe the cumulative probability of hallucinations and/or delusions over time. Participants will be determined to have met the primary endpoint if they have hallucinations and/or delusions on the basis of interview or initiate treatment with an antipsychotic medication.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No